CLINICAL TRIAL: NCT04355988
Title: Influence of Glycemic Levels on Healing of Periapical Lesions in Type 2 Diabetic Patients Following Primary Nonsurgical Root Canal Therapy
Brief Title: Glycemic Levels on Healing of Periapical Lesions in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Brhadyumna Bharath PGIDS
Record Dates: First submitted 2018-01-08; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2019-03

CONDITIONS: Periapical Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Well controlled diabetics (Active Comparator): Nonsurgical root canal treatment
  Interventions: Procedure: Nonsurgical root canal therapy
- Poorly controlled diabetics (Active Comparator): Nonsurgical root canal treatment
  Interventions: Procedure: Nonsurgical root canal therapy
- Healthy control group (Active Comparator): Nonsurgical root canal treatment
  Interventions: Procedure: Nonsurgical root canal therapy

INTERVENTIONS:
Procedure: Nonsurgical root canal therapy — After administration of LA and rubber dam isolation, acess cavity will be prepared using carbide burs in high speed hand piece with copious irrigation. Working length will be determined using root ZX apex locator and will be verified radiographically. Canal preparation will be done with protaper rotary instruments in which Sx to S2 will be used to shape the canals and F1 and F2 will be used to finish until the apex. 5ml of 5.25% NaOCl will be used as irrigant after each instrument. After instrumentation , the canals will be irrigated with 5.0 ml of 17% EDTA for 1minute followed by irrigation with 5.0 ml of 5.25% NaOCl. Canals will be dried with absorbent paper points, filled with calcium hydroxide paste and access cavity will be restored with IRM. Patients will be recalled after 1 week.At the next appointment, after paste removal, copious irrigation with 5.25% NaOCl will be done and canals will be dried with paper points. Canals will be obturated with Gutta-Percha and ZOE based sealer.
  Other Names: Root canal treatment

SUMMARY:
Increased incidence of peri-radicular lesions have been reported in diabetic patients which has been implicated due to compromised immune response. Much research has been done on the pathogenesis and progression of this lesion in diabetic patients. Although there are few studies which focus on healing of periradicular lesions after nonsurgical root canal treatment. There is a lacunae in literature which highlights peri-radicular healing after nonsurgical root canal treatment in relation to Glycaemic control in diabetic patients measured in terms of HbA1c levels.

DETAILED DESCRIPTION:
Diabetes mellitus is defined as a group of metabolic disorders characterized by chronic hyperglycemia with disturbances in carbohydrates, fat, and protein metabolism resulting from defects in insulin secretion, insulin action, or both. The effects of diabetes mellitus include long-term damage, dysfunction and failure of various organs: eyes, kidneys, nerves, heart, and blood vessels . Diabetes Mellitus is broadly classified into two types. Diabetes due to reduced insulin secretion from islet cells of pancreas is are known as type 1 and Diabetes due to combination of insulin resistance , reduced or increased insulin secretion are known as type 2.

One of the main detrimental effects of diabetes is its downregulation of immune system. It affects the immune cell function, up-regulates cytokines from monocytes or leukocytes and down-regulates the various growth factors predisposing to chronic inflammation, progressive tissue breakdown and reduced tissue repair capacity . So body becomes increasingly susceptible to infections and worsens if the blood glucose levels are not brought back to normal range .Oral symptoms of uncontrolled diabetes may comprise a plethora of conditions, such as dry mouth, tooth decay, periodontal diseases, delayed wound healing, and increased incidence of infection following surgery.

Diabetes mellitus inhibits collagen fibril formation and also interferes with collagen cross-linking and may impair degradation of matrix proteins and subsequent tissue remodeling , leading to poor wound healing in diabetics. Poor wound healing is similar in diabetic dental pulp.

Apical periodontitis is a chronic inflammatory lesion of the periapical region caused due to release of infectious products from the infected root canal system in the case of necrotic non vital pulp. It is characterized by periapical bone loss which does not heal unless the irritating agent is removed.

Thus, pro-inflammatory status and impaired immune response associated with systemic diseases can affect the reparative response of the dental pulp and periapical healing.Periapical immune response localizes the infection within the confines of the root canal system and prevents its systemic dissemination. In the host immune system, neutrophil is the first defense line when pathogens invade. Diabetes mellitus seriously impairs the function and bactericidal activity of neutrophils.

Apical periodontitis and chronic periodontitis share many common features including common microbiota and chronic nature of the disease. Several studies have been conducted linking periodontal disease and diabetes mellitus in terms of prevalence and worsening of glycaemic control in diabetic's patients.

Many studies have been done focusing on the effect of periodontal therapy on glycemic control in diabetes, including reviews and meta-analysis Although there are few studies which focus on healing of periradicular lesions after nonsurgical root canal treatment. Further research is necessary in this area to solidify our understanding on periapical healing and glycaemic control.

Aims and objectives To evaluate the clinical and radiographic success of primary non-surgical root canal treatment in teeth with apical periodontitis in good controlled/poor controlled diabetics To evaluate the clinical and radiographic success of primary non-surgical root canal treatment in teeth with apical periodontitis in diabetic patients (well controlled and poor controlled diabetics)/non-diabetics.

To evaluate the HbA1c levels as a means of glycemic control during the treatment of apical periodontitis in well controlled/poor controlled diabetic patients.

MATERIALS AND METHODS This study will be conducted in the department of conservative dentistry and endodontics, post graduate institute of dental sciences, Rohtak. Study subjects will be obtained from the pool of OPD patients in the Department of conservative dentistry and endodontics, PGIDS, Rohtak. Protocol for the study will be submitted for approval to institutional ethical committee of PGIDS Rohtak.

METHODOLOGY Prior to treatment a thorough clinical and radiological examination will be carried out.

A thorough history will be taken from each patient. Prior informed consent will be taken after explaining the procedure, risks and benefits.

Clinical procedure:

A total of 75 patients (n=25 in each group) will be included in the study

Sample size determination:

Sample size was determined using Karlsson's method with a power of 0.90 , P < 0,05% and standard deviation ± 0.50 according to which a sample of minimum 21 patients in each group was calculated , but keeping in mind the attrition a total of 25 patients will be recruited in each group .

First Appointment

Mature mandibular permanent molar with diagnosis of apical periodontitis (as confirmed clinically & by periapical radiograph) will be chosen for the study.

All periapical radiographs will be exposed by using constant kVP, mA and exposure time (70 KVP, 8 mA, 0.8 sec.) with a Rinn paralleling device and processed manually.

A customized zig will be prepared using addition silicone for each patient to keep as a future reference for film placement.

Fasting and post prandial blood glucose test & glycosylated hemoglobin (HbA1c) test will be done to evaluate the diabetic status of the patient.

Patients will be divide into three groups Good control diabetic patients- HbA1c levels ranging from 6.5%-7.5% Poor control diabetic patients-HbA1c levels greater than 7.5% Non diabetic Healthy controls-HbA1c levels less than 6.5% After administration of local anesthesia, rubber dam isolation of involved tooth will be done.

Acess cavity will be prepared using carbide burs in high speed hand piece with copious irrigation.

Negotiation of canals will be done. Working length will be determined using root ZX apex locator and will be verified radiographically.

Coronal enlargement will be done using Gates-Glidden drills. Hand files No. 10, 15 and 20 were used till working length (WL) to prepare a smooth reproducible glide path.

Canals will be prepared using the crown down technique with protaper rotary instruments in which coronal enlargement will be be done by Sx,S1 and S2. Finishing until the apex will be done by F1 and F2.

5ml of 5.25% sodium hypochlorite will be used for optimal irrigation after each instrument.

After completion of canal instrumentation , the canals will be irrigated with 5.0 ml of 17% ethylene-diamine-tetra acetic acid for 1minute followed by a final irrigation with 5.0 ml of 5.25% sodium hypochlorite Canals will be dried with absorbent paper points and filled with a paste of calcium hydroxide; the access cavity will be restored with intermediate restorative material.

The Patients will be recalled after 1 week. Second Appointment At the next appointment, the paste will be removed with H-files, copious irrigant with 5.25% NaOCl will be done; and canals will be dried with paper points.

Canals will be obturated with the Gutta-Percha and zinc Oxide-Eugenol based sealer.

After obturation, the cavity will be restored permanently. Immediate post-operative radiograph will be taken using preset exposure parameters and will be processed manually Follow up clinical and radiographic examination will be carried out at 3 months, 6 months, 9 months and 12th month.

ELIGIBILITY:
Inclusion Criteria-

1. Known patients of diabetes mellitus type 2 with HbA1c > 6.5%
2. Mature permanent mandibular posterior tooth having apical periodontitis
3. requiring primary root canal treatment
4. Age between 30 - 65 years.
5. A radiographic evidence of periapical radiolucency (minimum size ≥ 2mm×2mm) and a diagnosis of pulpal necrosis, as confirmed by negative response to cold and electrical tests; and absence of bleeding on entering the pulp chamber.

Exclusion Criteria-

1. Patient having advanced periodontal disease
2. Patient having systemic disorders other than diabetes
3. Pregnancy
4. Procedural errors
5. History of antibiotic intake in past one month

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Clinical Success | Baseline to one year
  Absence of signs and symptoms Absence of tenderness to percussion Tooth mobility of grade 1 or less Absence of associated soft tissue swelling or tenderness to palpation Attachment loss of less than 5mm .
  Two experienced observers with no knowledge of the treatment protocol will independently examine the immediate post obturation and follow up radiographs, mounted side by side, under controlled conditions. The treatment is considered successful only when both clinical and radiographic criteria are met. The worst outcome of an individual root decide the overall outcome for the tooth. In the event of disagreement, the two observers will meet to discuss their findings and came to an agreement.

SECONDARY OUTCOMES:
Radiographic success | Baseline to one year
  Absence of periapical alterations (radiolucency at furcal or periapical region) Scoring of each tooth will be done according to the following five point scale (PAI)
  Score Description
  1. Normal Periapical structure
  2. Small changes in bone structure
  3. Changes in bone structure with some mineral loss
  4. Periodontitis with well defined radiolucent area
  5. Severe periodontitis with exacerbating feature
  Lesions with a PAI score < 2 was considered

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No